CLINICAL TRIAL: NCT06295302
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIa Study to Explore the Efficacy, Safety, and Pharmacokinetic Profile of HWH486 in Adults With Chronic Spontaneous Urticaria(CSU)
Brief Title: A Study to Explore the Efficacy and Safety of HWH486 in Adults With Chronic Spontaneous Urticaria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Biological Medicine Industrial Technology Institute Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFCU-IIa-202308
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HWH486 (Experimental)
  Interventions: Drug: HWH486
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HWH486 — HWH486 capsule was administrated orally
  Arms: HWH486
Drug: Placebo — Matching placebo was administrated orally
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-bind and placebo-controlled phase IIa dose-finding study to assess the safety and efficacy of HWH486 in adults with chronic spontaneous urticaria (CSU). In addition, the pharmacokinetic characteristics will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤70 years old;
2. Participants with chronic spontaneous urticaria (CSU) at the time of randomization as defined by the following: presence of itch and hives for ≥ 6 consecutive weeks prior to screening, despite second generation H1-antihistamine during this period; Urticaria Activity Score (UAS7) (range 0-42) ≥16, Hives Severity Score (HSS7) (range 0-21) ≥ 6 and Itch Severity Score (ISS7) (range 0-21) ≥ 6 during 7 consecutive days prior to randomization; CSU duration ≥6 months prior to screening (defined as the onset of CSU as determined by the investigator based on all available supporting documentation).
3. Willing and able to complete the Urticaria Participant Daily eDiary (UPDD) for the duration of the study;
4. Willing to take background medication and emergency medication according to the study protocol.

6) Written informed consent signed voluntarily by the patient or their legal representatives.

Exclusion Criteria:

1. Previous use of HWH486 or other Bruton's tyrosine kinase(BTK) inhibitors;
2. Participants having a predominant or sole trigger of their chronic urticaria (chronic inducible urticaria);
3. Any other skin disease associated with chronic itching that might influence in the investigator's opinion the study evaluations and results, e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis
4. With symptoms or signs of progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, neurological, psychiatric, or brain disease, or with a history of gastrointestinal bleeding that is associated with a significant risk of bleeding or coagulopathy, or is clinically significant (such as requiring hospitalization or blood transfusion), or with other chronic medical conditions that are not eligible for participation in this clinical trial, or having a history of malignancy, other than non-metastatic basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of the cervix with appropriate treatment and no signs of recurrence;
5. Clinically important laboratory test indicators are abnormal, including: abnormal blood routine: hemoglobin (Hb) < 100g/L, or white blood cell count (WBC) < 3.5×10^9/L; Abnormal liver function: aspartate aminotransferase (AST) ≥1.5×ULN, or alanyl aminotransferase (ALT) ≥1.5×ULN, or total bilirubin (TBIL) ≥1.5×ULN; Abnormal renal function: creatinine (Cr) ≥1×ULN; any other laboratory test indicators that researchers think may affect the evaluation of test results;
6. Active and uncontrolled viral and bacterial infections at the time of screening, such as human immunodeficiency virus(HIV), hepatitis B virus(HBV), hepatitis C virus (HCV), syphilis, tuberculosis test results, or if there are any clinical symptoms of bacterial, viral, parasitic or fungal infection requiring treatment;
7. Pregnant or breastfeeding women; having pregnancy plans during the clinical trial and within 1 month after the last dose, and do not want to take medically accepted reliable contraceptive methods;
8. History of allergy to any investigational therapeutic drug or its excipients;
9. History or evidence of alcohol or drug abuse within the six months prior to randomization;
10. Use of other immunosuppressive drugs, including but not limited to hydroxychloroquine, methotrexate, cyclosporin A, cyclophosphamide, tacrolimus, mycophenolate, tripterygium, and compound glycyrrhizin, within 30 days or 5 half-lives (whichever is older) prior to screening;
11. The investigator determines that the subjects have any conditions that make them unfit to participate in the experiment (such as weak health, poor compliance, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Urticaria Activity Score (UAS) over a 7-day period (UAS7) | Baseline, Week 4
  Weekly Urticaria Activity Score (UAS7; range 0-42; higher scores reflect greater disease activity)

SECONDARY OUTCOMES:
Change in Hive Severity Score (HSS) over a 7-day period (HSS7) | Baseline to Week 4
  Weekly Hives Severity Score (HSS7; range 0-21; higher scores reflect greater wheals)
Change in Itch Severity Score (ISS) over a 7-day period (ISS7) | Baseline to Week 4
  Weekly Itch Severity Score (ISS7; range 0-21; higher scores reflect greater itching)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital,Sichuan University, Chengdu, Sichuan, China